CLINICAL TRIAL: NCT07248137
Title: Acute Effects of Different Physical Exercise Conditions in Patients With Peripheral Arterial Disease
Brief Title: Acute Effects of Exercise in Peripheral Arterial Disease Patients
Acronym: VESSEL-FIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University Miguel de Cervantes (Other)
Collaborators: Hospital Clínico Universitario de Valladolid. Angiology and Vascular Surgery Department. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PI-DOC009- VESSEL-FIT
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Aerobic Physical Exercise; Traditional Strength Exercise; Circuit Strength Exercise; Control
Keywords: Intermittent claudication; Proteomic markers; Vascular disease; Physiotherapy
MeSH Terms: conditions — Intermittent Claudication; Vascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The researcher responsible for analyzing the data will be blinded to the study conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic exercise (Experimental): Intermittent walking will be performed on a treadmill (F2W DUAL, BHFitness®, Spain). There will be 8 sets of 2 minutes in duration at an intensity equivalent to the level at which the patient experienced claudication symptoms. The recovery period between each set will be two minutes. All training sessions will conclude with a cool-down period of 5 minutes of walking at 50-60% of peak heart rate, followed by 3 minutes of joint mobility exercises. Throughout the session, heart rate will be continuously monitored using a heart rate monitor (Polar H10, Polar Electro Ltd., Kempele, Finland) and the Polar Team application (Polar Electro Ltd., Kempele, Finland).
  Interventions: Other: Aerobic exercise
- Traditional strength exercise (Experimental): Two sets will be performed with a moderate-to-high effort level (15-16 repetitions out of 20RM) consisting of 6 multi-joint exercises. The recovery period after each set will be two minutes of passive rest. Each participant will be asked to move the load as quickly as possible during each repetition. All training sessions will conclude with a cool-down period of 5 minutes of walking at 50-60% of peak heart rate, followed by 3 minutes of joint mobility exercises. Throughout the session, heart rate will be continuously monitored using a heart rate monitor (Polar H10, Polar Electro Ltd., Kempele, Finland) and the Polar Team application (Polar Electro Ltd., Kempele, Finland).
  Interventions: Other: Traditional strength exercise
- Circuit strength exercise (Experimental): Two sets (rounds) will be performed with a moderate-to-high effort level (15-16 repetitions out of 20RM) in a circuit consisting of 6 multi-joint exercises. The recovery time between exercises will be the minimum required to change exercises, and the recovery between sets (rounds) will be two minutes of passive rest. Each participant will be asked to move the load as quickly as possible during each repetition. All training sessions will conclude with a cool-down period of 5 minutes of walking at 50-60% of peak heart rate, followed by 3 minutes of joint mobility exercises. Throughout the session, heart rate will be continuously monitored using a heart rate monitor (Polar H10, Polar Electro Ltd., Kempele, Finland) and the Polar Team application (Polar Electro Ltd., Kempele, Finland).
  Interventions: Other: Circuit strength exercise
- Control (No Intervention): Control. No intervention

INTERVENTIONS:
Other: Aerobic exercise — Intermittent walking will be performed on a treadmill (F2W DUAL, BHFitness®, Spain). There will be 8 sets of 2 minutes in duration at an intensity equivalent to the level at which the patient experienced claudication symptoms. The recovery period between each set will be two minutes. All training sessions will conclude with a cool-down period of 5 minutes of walking at 50-60% of peak heart rate, followed by 3 minutes of joint mobility exercises. Throughout the session, heart rate will be continuously monitored using a heart rate monitor (Polar H10, Polar Electro Ltd., Kempele, Finland) and the Polar Team application (Polar Electro Ltd., Kempele, Finland).
  Arms: Aerobic exercise
Other: Traditional strength exercise — Two sets will be performed with a moderate-to-high effort level (15-16 repetitions out of 20RM) consisting of 6 multi-joint exercises. The recovery period after each set will be two minutes of passive rest. Each participant will be asked to move the load as quickly as possible during each repetition. All training sessions will conclude with a cool-down period of 5 minutes of walking at 50-60% of peak heart rate, followed by 3 minutes of joint mobility exercises. Throughout the session, heart rate will be continuously monitored using a heart rate monitor (Polar H10, Polar Electro Ltd., Kempele, Finland) and the Polar Team application (Polar Electro Ltd., Kempele, Finland).
  Arms: Traditional strength exercise
Other: Circuit strength exercise — Two sets (rounds) will be performed with a moderate-to-high effort level (15-16 repetitions out of 20RM) in a circuit consisting of 6 multi-joint exercises. The recovery time between exercises will be the minimum required to change exercises, and the recovery between sets (rounds) will be two minutes of passive rest. Each participant will be asked to move the load as quickly as possible during each repetition. All training sessions will conclude with a cool-down period of 5 minutes of walking at 50-60% of peak heart rate, followed by 3 minutes of joint mobility exercises. Throughout the session, heart rate will be continuously monitored using a heart rate monitor (Polar H10, Polar Electro Ltd., Kempele, Finland) and the Polar Team application (Polar Electro Ltd., Kempele, Finland).
  Arms: Circuit strength exercise

SUMMARY:
Peripheral arterial disease (PAD) affects over 200 million people worldwide and is caused by narrowing of the arteries. Intermittent claudication, characterized by pain when walking, is its main symptom. Despite the proven benefits of exercise, there is no optimal protocol for treatment. To analyze the effects of different exercise conditions on proteomic and physiological markers in patients with PAD and to determine their preferences regarding exercise conditions. A clinical cross-over study with four randomized experimental conditions (aerobic training, traditional strength training, circuit training and control) will be conducted. Patients with grade IIa-IIb PAD according to the Leriche-Le Fontaine scale will be recruited from the Department of Angiology and Vascular Surgery Department of the Hospital Clínico Universitario de Valladolid. In each experimental session, measurements of cardiorespiratory capacity, post-exercise oxygen debt, ankle-brachial index, blood flow, peripheral oxygen saturation, perceived exertion, heart rate variability and blood proteome changes will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Patients diagnosed with peripheral arterial disease at grade IIa or IIb according to the Leriche-Fontaine classification.

Exclusion Criteria:

* Patients with dementia or cognitive impairment.
* Patients with recent major surgery (≤12 months) or lower limb amputations.
* Patients institutionalized in healthcare facilities.
* Patients dependent on a wheelchair.
* Patients with any other condition contraindicating participation in an exercise program.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Blood Flow | Week 1 (baseline), Weeks 2-4 (15 minutes post-intervention)
  An ultrasound machine will be used to measure blood flow in the femoral artery, quantifying changes in the velocity and diameter of the artery in the lower extremity with the lowest ABI. Blood flow measurements will be conducted with the participant in a supine position. During the first experimental visit, the measurement site will be determined, where all measurements will take place. This measurement site corresponds to the common femoral artery, just below the inguinal ligament, and approximately 2 cm above the bifurcation into the superficial and deep femoral arteries.
Peripheral oxygen saturation | Week 1 (baseline), Weeks 2-4 (during each intervention session)
  Changes in peripheral oxygenation levels in the gastrocnemius will be evaluated during physical exercise. For this purpose, near-infrared spectroscopy (NIRS) will be used, which utilizes a wavelength of 700-900 nm to assess the concentration of oxygenated and deoxygenated hemoglobin and the total blood volume. The NIRS device MOXY Monitor (Moxy, Fortiori Design LLC, Minneapolis, MN, USA) will be used.
Heart rate variability | Week 1 (baseline), Weeks 2-4 (during intervention and 24, 48, and 72 hours post-intervention)
  By monitoring the heart rate of participants, heart rate variability (HRV) will be assessed, which reflects the variation in the time intervals between beats (R-R intervals) and serves as a useful tool for monitoring patient health, as it estimates the balance between the sympathetic and parasympathetic branches of the autonomic nervous system. To evaluate HRV, a Polar H10 heart rate monitor (Polar Electro Oy, Kempele, Finland) and a mobile application, specifically Elite HRV, will be used. Heart rate variability will be monitored daily during the week leading up to the initial assessment visits. Participants will be instructed to take the measurement for the first 5 minutes after waking up and while fasting.
Proteomics | Weeks 2-4 (5 minutes prior to exercise and 5 minutos post-intervention)
  A blood sample will be collected during the last 5 minutes of the pre-session and after completing the experimental condition, just before a 15-minute post-session rest. Venous blood will be drawn from the antecubital vein and stored at 4°C to prevent clotting and minimize protein degradation. Samples will be centrifuged at 1500 g for 10 minutes at 4°C, discarding the remaining sample. Ten microliters of protease inhibitor will be added to each 1.0 ml plasma aliquot, stored at -80°C for later analysis, with only one freeze-thaw cycle permitted. All samples will be prepared within 1 hour of collection and must show no hemolysis.
  Peptide identification will be performed using Proteome Discoverer (version 2.1.0.81) and SEQUEST-HT, analyzing data in the Uniprot database (January 25, 2024; 20,433 reviewed entries). Identified peptides with a false discovery rate (FDR) of 1% or less will quantify the relative abundance of each protein.

SECONDARY OUTCOMES:
Post-exercise oxygen debt | Weeks 2-4 (after every intervention session)
  Post-exercise oxygen debt (EPOC) will be calculated every minute for 12 minutes following the completion of exercise using the following formula: EPOC (L·min-¹) = post-exercise VO2 (L·min-¹) - resting VO2 (L·min-¹). Subsequently, EPOC will be converted into energy expenditure with the conversion of 1L of O2 = 4.64 kcal to exclude the rapid glycolytic resynthesis of adenosine triphosphate (ATP) as part of the conversion of O2 consumption into energy expenditure (EE).
Perceived exertion | Weeks 2-4 (right after every intervention session and 24, 48, and 72 hours post-intervention)
  During the four experimental conditions, perceived exertion will be monitored using the Rating of Perceived Exertion (RPE) scale. The RPE will be recorded after each set or circuit round. Immediately after completing the last set of each condition, participants will be asked to indicate their perceived exertion for the entire session.
  Scales go from 0 (no exertion) to 10 (maximal exertion possible).
Satisfaction with the type of training | Weeks 2-4 (right after every intervention session and 24 and 48 post-intervention)
  At the end of each session, satisfaction will be evaluated using a numerical scale from 0 to 10, where the highest score indicates maximum satisfaction with the type of training.

OTHER OUTCOMES:
Levels of physical activity. | Week 1 (baseline)
  Physical activity levels will be evaluated using the International Physical Activity Questionnaire (IPAQ), consisting of 7 questions for stratifying activity levels. Additionally, five GT3X+ accelerometers, updated to Firmware v1.9.2, will estimate physical activity. Each participant will wear the accelerometer securely on their right hip for one week, secured with an elastic belt. The ActiGraph GT3X+ (ActiGraph, Pensacola, Florida, USA) is lightweight (19 g), compact (4.6 × 3.3 × 1.5 cm), and features a rechargeable lithium polymer battery. It includes a solid-state triaxial accelerometer that collects data in three axes: vertical (Y), horizontal (X), and depth (Z). The device measures accelerations from -6 to 6 Gs and digitizes the output with a 12-bit analog-to-digital converter (ADC) at up to 100 Hz. The signal is filtered, and output is provided in "counts," reflecting the amplitude and frequency of movements over time.
Ankle-brachial index (ABI) | Week 1 (Baseline)
  A Doppler ultrasound machine with spectral wave analysis (Hadeco®) will be used to obtain systolic pressures in the right brachial artery, the dorsal artery of the foot, and the posterior tibial artery. To maximize accuracy, each pressure will be measured twice. The ankle-brachial index for each leg will be calculated by taking the ratio of the systolic pressure of the anterior or posterior tibial artery (whichever is higher) to the systolic pressure of the highest humeral artery (right or left). Normal values are considered to be 1.2-0.9 mmHg. A value above 1.2 mmHg will indicate arterial calcification, while a value below 0.9 mmHg will be considered pathological.
Cardiorespiratory capacity | Week 1 (baseline)
  The mean and peak values for gas exchange will be recorded in ml/kg·min. The gas analyzer used in this study is the Cortex Metalyzer 3B (Leipzig, Germany).
  A submaximal incremental treadmill walking test will be conducted under constant monitoring with a heart rate monitor and a portable gas analyzer. This test will be performed at a constant speed of 3.2 km/h, with 2% increases in incline at two-minute intervals. During the test, subjects will be asked to report the onset of the first symptoms of claudication.
Diastolic and systolic blood pressure | Week 1 (baseline), Weeks 2-4 (right before every intervention session and 24 hours post-intervention)
  For blood pressure measurement, an automatic Omron M3 blood pressure monitor (Omron Healthcare Co., Ltd., Kyoto, Japan) will be used. The participant should sit in a comfortable chair with lumbar support for at least 5 minutes before the measurement. They will be asked to place both feet flat on the floor, without crossing their legs, and rest the arm with the cuff on a table at chest height, with the palm facing up. Ensuring that the cuff is properly fitted but not too tight and in contact with bare skin, the blood pressure measurement will proceed. During this process, the subject should refrain from speaking to ensure an accurate and reliable reading. The obtained values will be recorded according to standard blood pressure measurement procedures. This protocol aims to ensure accurate and comfortable measurements to obtain reliable and consistent results in blood pressure evaluation.